CLINICAL TRIAL: NCT00842699
Title: Characterization of Immunological Profile of Renal Transplant Patients Undergoing Induction Treatment With Thymoglobulin vs. IL-2 Receptor Antagonist Basiliximab
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Nader Najafian, MD, Brigham and Women's Hospital
Other Study IDs: 2008p000774; Genzyme
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients receiving IL-2 receptor antagonist (Simulect) as induction treatment
- 2: patients receiving Thymoglobulin as induction treatment

SUMMARY:
The goal of the study is to find out the effects of two different drugs used at the beginning of organ transplantation on different populations of immune cells in the body of patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients considered for transplantation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: renal transplant recipients and living donors if available
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to look for expansion of regulatory T cells at one year. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nader Najafian, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States